CLINICAL TRIAL: NCT00238628
Title: A Phase I/II Study of Bexarotene in Combination With ZD 1839 (IRESSA) in the Third Line Treatment of Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Phase I/II Study of Bexarotene in Combination With ZD1839 (IRESSA®) in the Treatment of Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Ligand Pharmaceuticals (Industry); AstraZeneca (Industry)
Responsible Party: Charlotte D Jacobs, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUN0005; 80031; IRUSIRES0436; LUN0005; NCT00238628
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Bexarotene; Gefitinib

INTERVENTIONS:
Drug: Bexarotene
Drug: Iressa

SUMMARY:
The purpose of Phase 1 of this study is to evaluate the safety of the combination regimen, bexarotene and ZD1839. Phase II will evaluate the median survival, time to disease progression, and toxicity.

ELIGIBILITY:
Inclusion Criteria:- Patients must have histologically or cytologically confirmed NSCLC which is stage IIIB with malignant pleural effusion or stage IV and have failed therapy with at least a standard first line chemotherapy regimen, or be intolerant of standard chemotherapy.

* Patients may have non-measurable disease, or measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan).
* Patients with asymptomatic or treated brain metastases will be eligible if they last received therapy (including steroids) > 4 weeks from study entry and are felt to have a low likelihood of rapid deterioration from their brain metastases.
* Patients must have had at least 1 prior systemic therapy for NSCLC, or have shown intolerance to chemotherapy. Patients may not have received prior therapy with bexarotene, ZD1839, or erlotinib (Tarceva).
* At least 4 weeks must have elapsed from the time of major surgery and patients must have recovered from the effects of any significant procedure.
* A three week interval must have elapsed from the last dose of chemotherapy (30 days for investigational therapy), prior to beginning protocol therapy (6 weeks if nitrosoureas or mitomycin C). Palliative radiotherapy to bony sites of disease is allowed while on trial and up to time of enrollment provided patient has no significant side effects from the radiotherapy.
* Age >= 18 years.
* Life expectancy > 2 months.
* ECOG performance status 0-2.
* Women of childbearing potential must have a negative pregnancy test (serum ß HCG with a sensitivity of at least 50 mlU/L) within 7 days prior to initiation of treatment and must have used 2 reliable forms of effective contraception used simultaneously or have been sexually abstinent for at least 4 weeks prior to the negative pregnancy test through entry in the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  * Retinoid class agents are known teratogens.
* Female patients and male patients with female partners of childbearing potential must agree to sexual abstinence or to practice 2 reliable forms of effective contraception used simultaneously during the entire period of bexarotene capsule treatment and for at least 1 month after treatment is discontinued. Male patients must agree to use condoms if they have a female sexual partner who is, or may become, pregnant.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >= 3,000/ul
  * absolute neutrophil count >= 1,500/ul
  * platelets >= 100,000/ul
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <= 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR calculated creatinine clearance >= 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
  * triglycerides and cholesterol levels which are within normal limits or "normalized" with medication
* Patients may take the following agents, but with caution due to interactions with P450 metabolism: dexamethasone, protease inhibitors, ketoconazole and other azole antifungals, erythromycin and other macrolides antibiotics, grapefruit juice, other retinoid class drugs, beta-carotene compounds, and agents which enhance insulin secretion and sensitivity. They may not take phenytoin, carbamazepine, rifampicin, barbiturates, or St. John's Wort while on study.
* Ability to understand and the willingness to sign a written informed consent document Exclusion Criteria:- Insulin dependent diabetes
* Thyroid disease
* Patients may not have had chemotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study and must have recovered from adverse events due to agents administered more than 4 weeks earlier. Palliative radiotherapy is allowed to bony sites of disease.
* Patients may not be receiving any other investigational agents or have received any within 30 days prior to day 1 of study.
* Patients with known symptomatic brain metastases are excluded from this clinical trial because of their poor prognosis, those with treated, asymptomatic brain metastases are eligible proved they have not required any therapy including steroids for at least 4 weeks.
* Patients with a history of allergic reactions or sensitivity attributed to compounds of similar chemical or biologic composition to bexarotene and ZD1839 are excluded.
* Patients with triglycerides or cholesterol levels which are not within normal limits or "normalized" with medication will be excluded.
* Patients will be excluded for uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with another active malignancy except for non-melanoma skin cancers are excluded.
* Pregnant or breastfeeding women are excluded.
* Patients with risk factors for pancreatitis are excluded such as a history of pancreatitis, significant alcohol consumption or other factors which are deemed to put them at high risk.
* Patients taking systemic vitamin A in doses exceeding 15,000 IU/day within 14 days of study entry will be excluded.
* Patients who are unwilling to minimize exposure to ultraviolet light (sunlight) while on bexarotene will be excluded.
* Patients MAY NOT TAKE GEMFIBROZIL while on study due to interactions with bexarotene
* Patients may not take phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort while on the study.
* Patients with any evidence of clinically active interstitial lung disease will be excluded (patients with chronic stable radiographic changes who are asymptomatic need not be excluded)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2004-04; Primary Completion 2005-04 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Overall response rate (RECIST CRITERIA), time to progression, toxicity | Completed 9/2005
Pharmacokinetic analysis | Completed 12/2005
Median survival | Calculated Spring 2008
Overall response rate (RECIST CRITERIA), time to progression, toxicity | Final analysis Spring 2008

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte D Jacobs, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States